CLINICAL TRIAL: NCT01647815
Title: Ultrasound Comparison of the Surface of the Subclavian Vein (Arm in Abduction (90°) and External Rotation (90 °)) and the Surface of the Axillary Vein (Arms Along the Body) Versus the Surface of the Subclavian Vein (Arm Along the Body)
Brief Title: Ultrasound Comparison of the Surface of the Subclavian and the Axillary Vein Versus the Surface of the Subclavian Vein
Acronym: AnatoAbord
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LOCAL/2012/PJ-02; 2012-A00624-39 (Other: ANSM)
Record Dates: First submitted 2012-07-17; First posted 2012-07-24 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2015-03

CONDITIONS: Healthy Volunteers
Keywords: Axillary vein ultrasound; Subclavian vein ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 50 healthy volunteers (Experimental): The study population consists of healthy volunteers aged 18 to 50 years and without previous surgery, trauma, or thrombosis of the axilla or the shoulder girdle.
  Interventions: Procedure: Ultrasound measures

INTERVENTIONS:
Procedure: Ultrasound measures — Ultrasound will be used to measure the surfaces of the axillary and subclavian veins with the arms in different positions. Our goal is to compare the vein surface area available among different vein-position combinations. Our goal does not include testing specific devices.

SUMMARY:
The main objective of this study is the demonstration of an increase of over 50% of the surface visible on ultrasound (mm2) of the axillary vein and subclavian vein in arm abduction (90 °) and external rotation (90 °) with respect to the surface of the subclavian vein along the arm body.

DETAILED DESCRIPTION:
The secondary objective of this study is to investigate the anatomical relationships of these veins with the subclavian artery, the brachial plexus and the pleura, and assess the depth of the vein to the skin. Specifically, the following will be assessed:

* the depth of the vein (mm)
* the length of the minor axis (mm)
* the length of the major axis (mm)
* artery-vein distance (mm)
* vein-pleural distance (mm)
* the distance of the brachial plexus (mm)

ELIGIBILITY:
Inclusion Criteria:

* The volunteer must have given his/her informed and signed consent
* The volunteer must be insured or beneficiary of a health insurance plan
* The volunteer is 18 to 50 years old

Exclusion Criteria:

* The volunteer is participating in another study
* The volunteer is in an exclusion period determined by a previous study
* The volunteer is under judicial protection, under tutorship or curatorship
* The volunteer refuses to sign the consent
* It is impossible to correctly inform the volunteer
* The volunteer is pregnant, parturient, or breastfeeding
* The volunteer has a contraindication for the exams in this study
* Volunteer with a history of trauma or surgery in the axilla or the shoulder girdle
* Volunteer with a known history of venous thrombosis in the axillary and / or subclavian veins

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-08; Primary Completion 2012-08-10 (Actual); Study Completion 2012-08-10 (Actual)

PRIMARY OUTCOMES:
vein surface (mm^2), subclavian vein with arm along side the body | baseline (transversal); Day 0
vein surface (mm^2), subclavian vein with arm in abduction and external rotation | baseline (transversal); Day 0
vein surface (mm^2), axillary vein with arm along side the body | baseline (transversal); Day 0

SECONDARY OUTCOMES:
Vein depth (mm), subclavian vein with arms along side the body | baseline (transversal); Day 0
Length of minor axis (mm), subclavian vein with arms along side the body | baseline (transversal); Day 0
Length of major axis (mm), subclavian vein with arms along side the body | baseline (transversal); Day 0
Artery-vein distance is displayed in the section plane? yes/no | baseline (transversal); Day 0
  Ultrasound of subclavian vein with arm along side the body.
Artery-vein distance (mm) | baseline (transversal); Day 0
  Ultrasound of subclavian vein with arm along side the body.
  Artery-vein distance is displayed in the section plane? = yes
The vein-pleura distance is displayed in the section plane? yes/no | baseline (transversal); Day 0
  Ultrasound of subclavian vein with arm along side the body.
Vein-pleura distance (mm) | baseline (transversal); Day 0
  Ultrasound of subclavian vein with arm along side the body.
  The vein-pleura distance is displayed in the section plane? = yes
The distance to the brachial plexus is visualized in the sectional plane? yes/no | baseline (transversal); Day 0
  Ultrasound of subclavian vein with arm along side the body.
Distance to brachial plexus (mm) | baseline (transversal); Day 0
  Ultrasound of subclavian vein with arm along side the body.
  The distance of the brachial plexus is visualized in the sectional plane? = yes
Vein depth (mm), subclavian vein with arm in abduction and external rotation | baseline (transversal); Day 0
Length of minor axis (mm), subclavian vein with arm in abduction and external rotation | baseline (transversal); Day 0
Length of major axis (mm), subclavian vein with arm in abduction and external rotation | baseline (transversal); Day 0
Vein depth (mm), axillary vein with arm along side the body | baseline (transversal); Day 0
Length of minor axis (mm), axillary vein with arm along side the body | baseline (transversal); Day 0
Length of major axis (mm), axillary vein with arm along side the body | baseline (transversal); Day 0
Artery-vein distance is displayed in the section plane? yes/no | baseline (transversal); Day 0
  Ultrasound of subclavian vein with arm in abduction and external rotation.
Artery-vein distance (mm) | baseline (transversal); Day 0
  Ultrasound of subclavian vein with arm in abduction and external rotation.
  Artery-vein distance is displayed in the section plane? = yes
The vein-pleura distance is displayed in the section plane? yes/no | baseline (transversal); Day 0
  Ultrasound of subclavian vein with arm in abduction and external rotation.
The distance to the brachial plexus is visualized in the sectional plane? yes/no | baseline (transversal); Day 0
  Ultrasound of subclavian vein with arm in abduction and external rotation.
Vein-pleura distance (mm) | baseline (transversal); Day 0
  Ultrasound of subclavian vein with arm in abduction and external rotation.
  The vein-pleura distance is displayed in the section plane? = yes
Distance to brachial plexus (mm) | baseline (transversal); Day 0
  Ultrasound of subclavian vein with arm in abduction and external rotation.
  The distance of the brachial plexus is visualized in the sectional plane? = yes
Artery-vein distance is displayed in the section plane? yes/no | baseline (transversal); Day 0
  Ultrasound of axillary vein with arm along side the body.
Artery-vein distance (mm) | baseline (transversal); Day 0
  Ultrasound of axillary vein with arm along side the body.
  Artery-vein distance is displayed in the section plane? = yes
The vein-pleura distance is displayed in the section plane? yes/no | baseline (transversal); Day 0
  Ultrasound of axillary vein with arm along side the body.
Vein-pleura distance (mm) | baseline (transversal); Day 0
  Ultrasound of axillary vein with arm along side the body.
  The vein-pleura distance is displayed in the section plane? = yes
Distance to brachial plexus (mm) | baseline (transversal); Day 0
  Ultrasound of axillary vein with arm along side the body.
  The distance of the brachial plexus is visualized in the sectional plane? = yes
The distance to the brachial plexus is visualized in the sectional plane? yes/no | baseline (transversal); Day 0
  Ultrasound of axillary vein with arm along side the body.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Jeannes, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

REFERENCES:
- [Result] Sadek M, Roger C, Bastide S, Jeannes P, Solecki K, de Jong A, Buzancais G, Elotmani L, Ripart J, Lefrant JY, Bobbia X, Muller L. The Influence of Arm Positioning on Ultrasonic Visualization of the Subclavian Vein: An Anatomical Ultrasound Study in Healthy Volunteers. Anesth Analg. 2016 Jul;123(1):129-32. doi: 10.1213/ANE.0000000000001327. PMID 27149016
- [Derived] Roger C, Sadek M, Bastide S, Jeannes P, Muller L, Bobbia X, Lefrant JY. Comparison of the visualisation of the subclavian and axillary veins: An ultrasound study in healthy volunteers. Anaesth Crit Care Pain Med. 2017 Feb;36(1):65-68. doi: 10.1016/j.accpm.2016.05.007. Epub 2016 Aug 2. PMID 27495959